CLINICAL TRIAL: NCT00821639
Title: Reduction of Secondhand Smoke Exposure in Healthy Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Azam Baheiraei MPH,PhD/Principle Investigator, Tehran Univeristy of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: TUMS-6870
Record Dates: First submitted 2009-01-11; First posted 2009-01-13 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Secondhand Smoke Exposure
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Counseling, educational pamphlet and a sticker — Infants exposed to secondhand smoke will be recruited and randomized based on parents to receive or not receive counseling, an educational pamphlet and a sticker on SHS.

SUMMARY:
The purpose of this study is to assess the effects of a health center based counselling method for the prevention of infant exposure to secondhand smoke.

DETAILED DESCRIPTION:
This study, a two group randomised controled trial, investigates whether an intervention for parents would persuade them to enforce smoking bans inside the home and in other locations. A total of 130 parents with children aged 12 months or younger will be recruited. Each group (n=65) will complete a baseline and follow up questionnaire. Urine samples from the infants will be collected to measure the amount of cotinine, a metabolite of nicotine. The parent-report and infant's urinary cotinine measures will be obtained at baseline and at a 3-month follow up. In the intervention group, parents will be given three counselling sessions. For mothers, one being face to face and two telephone counselling and for fathers we will conduct three telephone counselling. The control group receives no intervention. Both groups will also complete a Fagerstrom test for nicotine dependence.

ELIGIBILITY:
Inclusion Criteria:

* Families with healthy infants under 12 months of age
* The infant resides with at least one smoking parent
* Parents being able to speak Persian and having a telephone

Exclusion Criteria:

* Parent(s) reporting consumption of other addictive substances
* Parent(s) in smoking cessation treatment

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Infant's urinary cotinine levels | At baseline and at a 3-month follow-up

SECONDARY OUTCOMES:
Home smoking bans status, Car smoking bans status, Parental cigarette consumption | At baseline and at a 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Azam Baheiraei, MPH, PhD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran